CLINICAL TRIAL: NCT02568293
Title: A Multicenter, Parallel, Blinded, Randomized Comparison of the Safety and Efficacy of Balloon Angioplasty Plus Intraluminal SBCV To Balloon Angioplasty Alone for Treatment of Stenosis or Occlusion Within the Femoropopliteal Artery
Brief Title: Angioplasty + SBCV vs. Angioplasty Alone for Femoropopliteal Artery Stenosis
Acronym: SHIELD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Symic Vascular (Industry)
Collaborators: Symic Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TP-1601
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBCV (Experimental): SBCV is administered to the site immediately post balloon dilation.
  Interventions: Other: SBCV
- Control (Placebo Comparator): Saline is used as a control and is delivered immediately post balloon dilation.
  Interventions: Other: Saline

INTERVENTIONS:
Other: SBCV — SBCV is a single use, sterile product that acts as a localized physical barrier at the vascular wall.
  Arms: SBCV
Other: Saline — Saline is used as a control.
  Arms: Control

SUMMARY:
The purpose of this study is to compare balloon angioplasty plus SBCV against balloon angioplasty alone for treatment of stenosis within the femoropopliteal artery.

DETAILED DESCRIPTION:
This first-in-human study will evaluate the safety and effectiveness of a novel adjunctive therapy, SBCV, used with balloon angioplasty as compared to balloon angioplasty plus a control agent (saline) when used for the treatment of stenosis within the femoropopliteal artery. Effectiveness will be measured by late lumen loss at 24 weeks post treatment as evaluated by an independent, blinded core lab.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for balloon angioplasty for stenosis of femoropopliteal lesion(s)
* Rutherford Clinical Category 1-4 (claudication or critical limb ischemia)
* Lesions are ≥70% stenosis by visual estimate
* A patent inflow artery free from significant lesion
* At least one patent native outflow artery to the ankle

Exclusion Criteria:

* History of haemorrhagic stroke within 3 months of screening
* History of myocardial infarction, thrombolysis or angina within 2 weeks of screening
* Renal failure or chronic kidney disease
* Severe calcification that renders the lesion undilatable

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | through 24 weeks
  The composite of no all-cause perioperative (≤30 day) mortality and none of the following events at 24 weeks following treatment:
  * Index limb amputation (above or below the ankle)
  * Index limb re-intervention
  * Index-limb-related death
Late Lumen Loss | 24 weeks
  LLL is defined as the difference between the minimum lumen diameter (MLD) immediately post-primary procedure and the MLD at follow-up as measured by an independent, blinded core lab.

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (7):
  - Royal Prince Alfred Hospital, Melbourne, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Flinders Medical Center, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Auckland City Hospital, Auckland, New Zealand